CLINICAL TRIAL: NCT07111442
Title: Fractional Flow Reserve-guided Percutaneous Renal Artery Stenting Versus Sham Procedure In Atherosclerosis Renal-vascular Hypertension Patients: a Double-blinded Multicenter Randomized Placebo-control Trial
Brief Title: A Placebo-controlled Trial of Fractional Flow Reserve-guided Percutaneous Renal Artery Stenting Among Atherosclerosis Renal-vascular Hypertension Patients
Acronym: FAIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022CR77V3.0
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Renal Artery Stenosis Atherosclerotic; Secondary Hypertension Renal Arterial
MeSH Terms: interventions — Dopamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Registry group (Other): If FFR ≥ 0.80, no renal artery stenting will be performed.
  Interventions: Diagnostic Test: renal artery fractional flow reserve measurement; Drug: dopamine
- Stenting group (Experimental): If FFR < 0.80, participants will be randomized in a 1:1 ratio to one of the following two intervention arms: Stenting Group: Renal artery tenting
  Interventions: Diagnostic Test: renal artery fractional flow reserve measurement; Drug: dopamine; Device: renal artery stent
- Control Group (Sham Comparator): If FFR < 0.80, participants will be randomized in a 1:1 ratio to one of the following two intervention arms: Control Group: Sham procedure
  Interventions: Diagnostic Test: renal artery fractional flow reserve measurement; Drug: dopamine; Other: sham stenting

INTERVENTIONS:
Diagnostic Test: renal artery fractional flow reserve measurement — Eligible participants who meet all inclusion and exclusion criteria will undergo renal angiography. On the day of angiography, a functional assessment of renal artery stenosis will be performed according to the Standard Operating Procedure (SOP) using a pressure wire under dopamine-induced maximal hyperemia to measure the Fractional Flow Reserve (FFR).
Drug: dopamine — Administer dopamine at 50 µg/kg via the renal artery to induce hyperemic.
Device: renal artery stent — Stent will be treated for the stenotic renal artery for patients randomized to stenting group
  Arms: Stenting group
Other: sham stenting — For participants randomized to the sham procedure, the procedure will last at least 15 minutes to simulate actual intervention according to SOP guidelines.
  Arms: Control Group

SUMMARY:
Objective: To determine whether percutaneous renal artery stenting guided by fractional flow reserve (FFR), in addition to standard medical therapy, provides superior therapeutic efficacy compared to medical therapy alone in patients with atherosclerotic renal artery stenosis and hypertension.

Study Design: A double-blind, multicenter, prospective, randomized, placebo-controlled (sham procedure) trial.

Primary Endpoint: The percentage reduction in daytime mean systolic blood pressure measured by ambulatory blood pressure monitoring (ABPM) from baseline to 3 months after the procedure.

Study Population: A total of 200 patients who are potential candidates for renal artery intervention will be enrolled. Participants must meet all of the following inclusion criteria to be eligible for the study.

Participant Screening and Enrollment: Once a patient is preliminarily assessed in the outpatient clinic and meets the clinical inclusion/exclusion criteria, written informed consent will be obtained, and the patient will enter a 1-week screening period. During this period, patients will perform home blood pressure monitoring using a calibrated Bluetooth-enabled device provided by the study team, which automatically uploads data. In addition, antihypertensive medications will be standardized to optimize blood pressure management.

If home BP measurements during the screening period continue to meet inclusion criteria, baseline ABPM will be conducted.

Following standardized renal angiography, patients whose renal anatomy meets the angiographic inclusion/exclusion criteria will undergo functional assessment of the stenotic lesion using a pressure wire and measurement of renal fractional flow reserve (FFR) under dopamine-induced maximal hyperemia, in accordance with the Standard Operating Procedure (SOP).

Patients who qualify will then be randomized based on FFR results using an Interactive Response Technology (IRT) system. All eligible patients will be assigned a unique subject identification number during screening, and randomization will occur on the day of angiography, ensuring allocation concealment and unbiased group assignment.

Study Intervention: Eligible participants who meet all inclusion and exclusion criteria will undergo renal angiography. On the day of angiography, a functional assessment of renal artery stenosis will be performed according to the Standard Operating Procedure (SOP) using a pressure wire under dopamine-induced maximal hyperemia to measure the Fractional Flow Reserve (FFR).

* If FFR ≥ 0.80, no renal artery stenting will be performed.
* If FFR < 0.80, participants will be randomized in a 1:1 ratio to one of the following two intervention arms:

  * Stenting Group: Renal artery stenting
  * Control Group: Sham procedure The randomization assignment will be blinded to participants and follow-up investigators. Only designated study investigators and the operating team will be aware of the group allocation. For participants randomized to the sham procedure, the procedure will last at least 15 minutes to simulate actual intervention according to SOP guidelines. Group allocation will remain blinded until the primary endpoint is assessed at 3 months post-procedure.

All participants, regardless of group assignment, will receive guideline-directed optimized medical therapy throughout the study period.

Study Duration and Follow-up: Participants will be followed for a total of 12 months with study visits scheduled at the following time points:

* 4 weeks post-procedure (telephone visit)
* 12 weeks (clinic visit)
* 6 months (clinic visit)
* 12 months (clinic visit)

To minimize the impact of antihypertensive medication adjustments on statistical outcomes, it is strongly recommended that no changes be made to antihypertensive regimens during the first 3 months after enrollment unless clinically necessary, such as in cases of:

* Systolic BP < 100 mmHg, or
* Systolic BP > 180 mmHg and/or diastolic BP > 100 mmHg. All changes to antihypertensive therapy (including drug type and dosage) will be documented in detail.

To ensure consistency and quality, standardized recommendations for antihypertensive drug selection and adjustment will be provided in accordance with current hypertension management guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older.
2. Documented history of hypertension and currently taking two or more antihypertensive medications with uncontrolled blood pressure (defined as daytime systolic BP ≥135 mmHg and/or diastolic BP ≥85 mmHg on optimized medication therapy, as measured by baseline ABPM).
3. Clinical evidence suggestive of renal artery stenosis, and scheduled for renal angiography.
4. Willing and able to provide written informed consent prior to initiation of any study-related procedures, and willing to comply with all study requirements.
5. Renal angiography shows ≥70% to <99% stenosis in at least one main renal artery with a reference vessel diameter of ≥4.0 mm.

Exclusion Criteria:

1. Systolic BP ≥200 mmHg and/or diastolic BP ≥120 mmHg on the day of randomization.
2. Suspected non-atherosclerotic causes of RAS, such as fibromuscular dysplasia or large-vessel vasculitis.
3. Pregnant or breastfeeding women.
4. Participation in another clinical trial that, in the investigator's opinion, could interfere with this study.
5. Stroke or TIA within 3 months and known ≥70% carotid artery stenosis.
6. Major surgery, myocardial infarction, or any interventional procedure within the past 30 days.
7. Known LVEF <30%.
8. Life expectancy ≤1 year.
9. Known allergy to contrast media or to any of the following medications: aspirin, clopidogrel.
10. History of renal transplantation.
11. Prior renal artery stenting or bypass surgery.
12. Affected kidney length <8 cm on Doppler ultrasound.
13. Serum creatinine >3.0 mg/dL (265.2 μmol/L) at baseline visit (measured by local laboratory).
14. Reference vessel diameter <4 mm or >8 mm on angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
The percentage reduction in daytime mean systolic blood pressure measured by ambulatory blood pressure monitoring from baseline to 3 months post-procedure. | from baseline to three months after procedure

SECONDARY OUTCOMES:
Percentage change in the composite index of antihypertensive medication use | from baseline to 3 months post-procedure
Percentage reduction in 24-hour/daytime/nighttime mean systolic blood pressure measured by ambulatory blood pressure monitoring | from baseline to 3 months post-procedure
Percentage reduction in systolic blood pressure measured by home blood pressure monitoring | from baseline to 3 months post-procedure
Percentage reduction in office systolic blood pressure | from baseline to 3 months post-procedure
Change in the number of antihypertensive medications | from baseline to 3 months post-procedure
Number of hypertensive emergencies | from baseline to 3 months post-procedure
Percentage reduction in daytime mean systolic blood pressure by ambulatory blood pressure monitoring | from baseline to 6 months post-procedure
Percentage reduction in daytime mean systolic blood pressure by ambulatory blood pressure monitoring | from baseline to 12 months post-procedure

OTHER OUTCOMES:
All-cause mortality | 1 year post-procedure
Cardiovascular death | 1 year post-procedure
Acute myocardial infarction | 1 year post-procedure
Non-fatal stroke | 1 year post-procedure
Rehospitalization for congestive heart failure | 1 year post-procedure
Progression of renal insufficiency (change in eGFR) or need for dialysis | 1 year post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided